CLINICAL TRIAL: NCT04171596
Title: Feasibility of Care Coordination in an Integrative Primary Care Concierge Practice
Brief Title: Feasibility of Care Coordination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00087885
Record Dates: First submitted 2019-11-19; First posted 2019-11-21 (Actual); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Care Coordination in Primary Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Primary care coordination (Experimental)
  Interventions: Behavioral: Primary care coordination

INTERVENTIONS:
Behavioral: Primary care coordination — A registered nurse currently employed at Duke Integrative Medicine, who is also trained as an integrative health coach, will serve in the PCC role. The intervention will flow as follows:
  The PCC will call study participants every 2 months during the 6 months (more frequently as needed) for a semi-structured phone check-in, and will track the intervention through the REDCap database. The PCC will use guiding questions to frame the call, but will also:
  Respond Ask follow-up questions Provide suggestions that are guided by the patient response and appropriateness to the individual situation and needs and scope of practice.
  Prior to the call, the PCC will review the patient chart to see if any outstanding orders, medical visits due, and review the patient health goals (known as the "pre-work").
  The PCC will call the patient to provide intervention. If patient is not available, the PCC will leave a message, or contact via MyChart to see about scheduling a time to talk.

SUMMARY:
The primary aim of this study is to determine feasibility of incorporating a primary care coordinator (PCC) into an integrative concierge primary care practice. Secondary aims include:

1. To determine whether the PCC intervention increases patient satisfaction and/or patient activation.
2. To determine whether regular telephone contacts from a PCC over a period of 6 months increases the number of visits and services by DIPC members.

DETAILED DESCRIPTION:
The Duke Integrative Primary Care (DIPC) clinic in Durham, North Carolina currently serves over 600 patients, and offers a full range of primary care services. The practice is a fee-based model where patients pay a monthly fee to access primary care services, and includes several membership benefits. These benefits include longer appointment times, visits with physicians trained in integrative medicine, access to the Duke Health and Fitness Center, on-site discounts, and use of facilities at Duke Integrative Medicine.

Preliminary information gathered show that DIPC members state reasons of value, cost and underutilization for cancelling their memberships. Underutilized primary care memberships may represent missed opportunities to increase patient satisfaction, improve patient outcomes, and maximize clinic revenue.

DIPC employs an administrative coordinator responsible for assisting patients with enrolling and renewing their primary care memberships, but to date, there has not been a clinical care coordinator role in the DIPC clinic.

This study will provide the basis for understanding the feasibility of incorporating care coordination into the Duke Integrative Primary Care practice. In addition, cost and effort of the care coordinator will be compared to additional volume, revenue and patient satisfaction data to increase understanding of the value proposition. Further, information gathered during this study could suggest possible impact on membership retention rates, as well as inform next steps for continuous improvement initiatives for the integrative primary care practice.

Primary aim: To determine feasibility of incorporating a PCC into an integrative concierge primary care practice.

Secondary aims:

1. To determine whether the PCC intervention increases patient satisfaction and/or patient activation.
2. To determine whether regular telephone contacts from a PCC over a period of 6 months increases the number of visits and services by DIPC members.

After each subject completes an online consent and a pre-intervention questionnaire housed in a REDCap database, the PCC intervention will begin for that subject. A registered nurse currently employed at Duke Integrative Medicine, who is also trained as an integrative health coach, will serve in the PCC role. The intervention will flow as follows:

The PCC will call study participants every 2 months during the 6 months (more frequently as needed) for a semi-structured phone check-in, and will track the intervention through the REDCap database. The PCC will use guiding questions to frame the call, but will also:

Respond Ask follow-up questions Provide suggestions that are guided by the patient response and appropriateness to the individual situation and needs and scope of practice.

Prior to the call, the PCC will review the patient chart to see if any outstanding orders, medical visits due, and review the patient health goals (known as the "pre-work").

The PCC will call the patient to provide intervention. If patient is not available, the PCC will leave a message, or contact via MyChart to see about scheduling a time to talk.

After the 6-month intervention is complete, the study coordinator will send each individual subject a link to the post-intervention questionnaire in REDCap, and will follow up with each subject to ensure completion of this questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Member of the Duke Integrative Primary Care clinic in Durham, NC who have been members for at least 1 year.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-02-14 (Actual); Primary Completion 2018-10-11 (Actual); Study Completion 2019-04-11 (Actual)

PRIMARY OUTCOMES:
Number of patients enrolled | 6 months
  Number of patients enrolled as measured by enrollment logs
Number of patients that completed minimum intervention | Up to 1 year
  Number of patients that completed a minimum of 3 intervention calls as measured by call logs

SECONDARY OUTCOMES:
Patient satisfaction | Up to 1 year
  Number of patients that stated they were satisfied as measured by an internally-designed questionnaire
Number of additional clinic visits | Up to 1 year
  Number of additional clinic visits as determined by visits scheduled due to referrals that happened within the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Glass, PhD, Principal Investigator — Duke University
Locations (1):
- Duke Integrative Medicine, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No